CLINICAL TRIAL: NCT02026856
Title: Therapeutic Effect of Sodium Selenite on Oxidative Stress in Patients With Severe Sepsis
Acronym: Se-AOX
Status: Completed | Type: Observational
Sponsor: Pavol Jozef Safarik University (Other)
Responsible Party: Principal Investigator, Kočan Ladislav, MD PhD, Pavol Jozef Safarik University
Other Study IDs: Se-AOX 109/2011
Record Dates: First submitted 2013-12-31; First posted 2014-01-03 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2013-12

CONDITIONS: Severe Sepsis
Keywords: oxidative stress, sepsis, selenium
MeSH Terms: conditions — Sepsis | interventions — Sodium Selenite

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Se-OI> 200: patients who received form of sodium selenite pentahydrate at 750 mg/day for 6 days immediately after admission to our department (1000 mg of sodium selenite pentahydrate = 333 micrograms of selenium) and oxygenation index (OI) by PaO2/FiO2 (partial pressure of oxygen in arterial blood/ fraction of inspired oxygen) was higher than 200
  Interventions: Drug: sodium selenite pentahydrate
- Se-OI <200: patients who received form of sodium selenite pentahydrate at 750 mg/day for 6 days immediately after admission to our department (1000 mg of sodium selenite pentahydrate = 333 micrograms of selenium) and oxygenation index (OI) by PaO2/FiO2 (partial pressure of oxygen in arterial blood/ fraction of inspired oxygen) was lower than 200
  Interventions: Drug: sodium selenite pentahydrate
- Placebo-OI> 200: patients who received continuous saline NaCl 50 ml/day for 6 days as a continuous infusion (excluding additional infusion therapy) and oxygenation index (OI) by PaO2/FiO2 (partial pressure of oxygen in arterial blood/ fraction of inspired oxygen) was higher than 200
  Interventions: Other: placebo - continuous saline NaCl 50 ml
- Placebo-OI <200: patients who who received continuous saline NaCl 50 ml/day for 6 days as a continuous infusion (excluding additional infusion therapy) and oxygenation index (OI) by PaO2/FiO2 (partial pressure of oxygen in arterial blood/ fraction of inspired oxygen) was lower than 200
  Interventions: Other: placebo - continuous saline NaCl 50 ml

INTERVENTIONS:
Drug: sodium selenite pentahydrate
  Groups: Se-OI <200; Se-OI> 200
Other: placebo - continuous saline NaCl 50 ml
  Groups: Placebo-OI <200; Placebo-OI> 200

SUMMARY:
This study looked at parenteral administration of selenium to septic patients and subsequently monitored dynamic changes of selected activities of antioxidant enzymes and the development of clinical status.

DETAILED DESCRIPTION:
Patients will be divided into two groups. Se-group who received selenium supplementation during hospitalization in the form of sodium selenite pentahydrate at 750 mg/day for 6 days immediately after admission to our department (1000 mg of sodium selenite pentahydrate = 333 micrograms of selenium) (Selenase, Vivax; selenium hereinafter).

The placebo group will receive continuous saline NaCl 50 ml/day for 6 days as a continuous infusion (excluding additional infusion therapy). Patients will be further divided into subgroups according to OI on the day of admission to ICU. The oxygenation index (OI) PaO2/FiO2 (partial pressure of oxygen in arterial blood/ fraction of inspired oxygen) ratio in patients will be calculated daily.

The determination of biochemical and hematological parameters of blood samples will be as a part of the routine diagnostic methods. Data collection for the Se-AOX study will be performed at two-day intervals: T1 (1st-2nd day), T2 (3rd-4th day) and T3 (5th-6th day). Kinetic methods for estimating the activities of glutathione peroxidase (GPx, E.C. 1.11.1.9), glutathione reductase (GR, E.C.1.6.4.2) will be performed using a kit (Sigma-Aldrich, Germany) and that of superoxide dismutase (SOD, E.C. 1.15.1.1) by means of the SOD-Assay Kit-WST (Fluka, Japan) following the user manual provided.

ELIGIBILITY:
Inclusion Criteria:

* sepsis, severe sepsis or septic shock, APACHE II score between 19 and 24 points after admission

Exclusion Criteria:

* mechanical ventilation for less than 24h, neuromuscular disease and terminal illness were also excluding criteria

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with APACHE II score between 19 and 24 points after admission with sepsis, severe sepsis or septic shock during hospitalization as defined by the International Sepsis Definitions Conference
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
mortality | 2 years

SECONDARY OUTCOMES:
The oxygenation index | 2 years
  PaO2/FiO2 (partial pressure of oxygen in arterial blood/ fraction of inspired oxygen)

OTHER OUTCOMES:
antioxidant enzymes | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- 1st clinic of anesthesiology and intesive care, University hospital of Louis Pasteur, Košice, Slovakia

REFERENCES:
- [Background] Kocan L, Vaskova J, Vasko L, Lakyova L, Kocanova H, Simonova J, Simon R, Firment J. [Acute multiple organ failure after endoscopic polypectomy]. Cas Lek Cesk. 2012;151(12):568-72. Slovak. PMID 23387814
- [Result] Kocan L, Firment J, Simonova J, Vaskova J, Guzy J. [Selenium supplementation in patients with severe acute pancreatitis]. Rozhl Chir. 2010 Aug;89(8):518-21. Slovak. PMID 21121149
- [Derived] Kocan L, Firment J, Pirnikova I, Farkasova Iannaccone S, Rybar D, Gnorikova J, Korcek J, Kocanova H, Torok P, Rapcanova S, Vaskova J. Full recovery of lung tissue after severe viral pneumonia H1N1: A case report with 10 years follow-up. Medicine (Baltimore). 2023 Feb 22;102(8):e33052. doi: 10.1097/MD.0000000000033052. PMID 36827018
- [Derived] Kocan L, Vaskova J, Vasko L, Simonova J, Simon R, Firment J. Selenium adjuvant therapy in septic patients selected according to Carrico index. Clin Biochem. 2014 Oct;47(15):44-50. doi: 10.1016/j.clinbiochem.2014.07.004. Epub 2014 Jul 12. PMID 25020262